CLINICAL TRIAL: NCT02662634
Title: A Safety and Feasibility Study of AGS-003-LNG for the Treatment of Stage 3 Non Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: GU Research Network, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGS-003-024
Record Dates: First submitted 2016-01-12; First posted 2016-01-25 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; resectable; non-small cell lung cancer; immunotherapy; autologous; dendritic cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed; Cisplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequential, no radiation (Experimental): AGS-003-LNG initiated after completion of platinum doublet chemotherapy. AGS-003-LNG induction = 1 dose administered every 3 weeks for 5 doses. Booster doses will then be administered every 12 weeks. A dose of AGS-003-LNG consists of (1.2 x 10-7 Dendritic cells.) Platinum-doublet chemotherapy can be any of the following determined by PI
  Carboplatin/Abraxane:
  ABRAXANE is 100 mg/m2 i.v. over 30 minutes on Days 1, 8, & 15 of each 21-day cycle; carboplatin Area Under Curve (AUC) 6 (C&G) on Day 1 of each 21-day cycle immediately after ABRAXANE.
  Carboplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day cycle in combination with carboplatin AUC 6 (C&G) i.v. 30 minutes after ALIMTA.
  Cisplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day with cisplatin 75 mg/m2 i.v., 30 minutes after ALIMTA.
  Carboplatin/Taxol TAXOL administered i.v. over 24 hrs at a dose of 135 mg/m2 followed by carboplatin, AUC 6 (C&G).
  Interventions: Biological: AGS-003-LNG; Drug: Carboplatin; Drug: Abraxane; Drug: Alimta; Drug: Cisplatin; Drug: Taxol; Radiation: Radiation Therapy
- Concurrent, no radiation (Experimental): AGS-003-LNG dosing initiated concurrently or subsequent to 3rd cycle of platinum doublet chemotherapy & radiation therapy. AGS-003-LNG induction = 1 dose administered every 3 wks for 5 doses. Booster doses will then be administered every 12 wks. A dose of AGS-003-LNG =1.2 x 10-7 Dendritic cells.
  Platinum-doublet chemotherapy can be any of the following determined by PI
  Carboplatin/Abraxane:
  ABRAXANE is 100 mg/m2 i.v. over 30 minutes on Days 1, 8, & 15 of each 21-day cycle; carboplatin AUC 6 (C&G) on Day 1 of each 21-day cycle immediately after ABRAXANE.
  Carboplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day cycle in combination with carboplatin AUC 6 (C&G) i.v. 30 minutes after ALIMTA.
  Cisplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day with cisplatin 75 mg/m2 i.v., 30 minutes after ALIMTA.
  Carboplatin/Taxol TAXOL administered i.v. over 24 hrs at a dose of 135 mg/m2 followed by carboplatin, AUC 6 (C&G).
  Interventions: Biological: AGS-003-LNG; Drug: Carboplatin; Drug: Abraxane; Drug: Alimta; Drug: Cisplatin; Drug: Taxol; Radiation: Radiation Therapy
- Sequential, radiation (Experimental): AGS-003-LNG initiated after completion of platinum doublet chemotherapy. AGS-003-LNG induction = 1 dose administered every 3 weeks for 5 doses. Booster doses will then be administered every 12 weeks. A dose of AGS-003-LNG consists of (1.2 x 10-7 Dendritic cells.) Platinum-doublet chemotherapy can be any of the following determined by PI
  Carboplatin/Abraxane:
  ABRAXANE is 100 mg/m2 i.v. over 30 minutes on Days 1, 8, & 15 of each 21-day cycle; carboplatin AUC 6 (C&G) on Day 1 of each 21-day cycle immediately after ABRAXANE.
  Carboplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day cycle in combination with carboplatin AUC 6 (C&G) i.v. 30 minutes after ALIMTA.
  Cisplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day with cisplatin 75 mg/m2 i.v., 30 minutes after ALIMTA.
  Carboplatin/Taxol TAXOL administered i.v. over 24 hrs at a dose of 135 mg/m2 followed by carboplatin, AUC 6 (C&G).
  Radiation therapy per PI
  Interventions: Biological: AGS-003-LNG; Drug: Carboplatin; Drug: Abraxane; Drug: Alimta; Drug: Cisplatin; Drug: Taxol; Radiation: Radiation Therapy
- Concurrent, radiation (Experimental): AGS-003-LNG dosing initiated concurrently during or subsequent to the 3rd cycle (3-week cycle) of platinum doublet chemotherapy & radiation therapy. AGS-003-LNG induction = 1 dose administered every 3 wks for 5 doses. Booster doses administered every 12 wks. A dose of AGS-003-LNG =1.2 x 10-7 Dendritic cells.
  Platinum-doublet chemotherapy choice of the following determined by PI
  Carboplatin/Abraxane:
  ABRAXANE is 100 mg/m2 i.v. over 30 minutes on Days 1, 8, & 15 of each 21-day cycle; carboplatin AUC 6 (C&G) on Day 1 of each 21-day cycle immediately after ABRAXANE.
  Carboplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day cycle in combination with carboplatin AUC 6 (C&G) i.v. 30 minutes after ALIMTA.
  Cisplatin/Alimta ALIMTA is 500 mg/m2 i.v. on Day 1 of each 21-day with cisplatin 75 mg/m2 i.v., 30 minutes after ALIMTA.
  Carboplatin/Taxol TAXOL administered i.v. over 24 hrs at a dose of 135 mg/m2 followed by carboplatin, AUC 6 (C&G).
  Radiation therapy per PI.
  Interventions: Biological: AGS-003-LNG; Drug: Carboplatin; Drug: Abraxane; Drug: Alimta; Drug: Cisplatin; Drug: Taxol; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: AGS-003-LNG — autologous dendritic cell immunotherapy
Drug: Carboplatin — Carboplatin is an anticancer drug ("antineoplastic" or "cytotoxic") chemotherapy drug. Carboplatin is classified as an "alkylating agent."
  Other Names: Paraplatin
Drug: Abraxane — Paclitaxel destroys cancer cells by preventing the normal breakdown of microtubules during cell division.
  Other Names: Protein-bound paclitaxel; nano-particle albumin-bound paclitaxel; nab-paclitaxel
Drug: Alimta — By inhibiting the formation of precursor purine and pyrimidine nucleotides, pemetrexed prevents the formation of DNA and RNA, which are required for the growth and survival of both normal cells and cancer cell
  Other Names: Pemetrexed
Drug: Cisplatin — Binds to and causes crosslinking of DNA, which ultimately triggers apoptosis
  Other Names: Cisplatinum; platamin; neoplatin; cismaplat; cis-diamminedichloroplatinum(II)
Drug: Taxol — Mechanism of action involves interference with the normal breakdown of microtubules during cell division.
  Other Names: Paclitaxel
Radiation: Radiation Therapy — Causes DNA strand breaks.

SUMMARY:
Feasibility and Safety study of autologous dendritic cell immunotherapy (AGS-003-LNG) in patients with resectable non-small cell lung cancer.

DETAILED DESCRIPTION:
Feasibility and Safety study of autologous dendritic cell immunotherapy (AGS-003-LNG) in patients with resectable non-small cell lung cancer. Non-small cell lung cancer tumor will be resected from the patient. RNA from the tumor will be amplified and subsequently electroporated into matured, autologous dendritic cells. The dendritic cells with tumor RNA will be dosed back to the patient. Study will investigate feasibility and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years.
2. Newly diagnosed non-small cell lung cancer indicated for routine lobectomy, mediastinoscopy, wedge resection, thoracotomy or Video-assisted thoracoscopic surgery (VATS) procedures with tumor collection.
3. Stage III (T1-3, N1-2, M0) of any histology.
4. Scheduled for routine lobectomy, mediastinoscopy, wedge resection, thoracotomy or VATS procedures.
5. Signed and dated informed consent document for study participation.

After tumor collection, potential subjects must meet all the following criteria to be enrolled in study treatment:

1. Successful RNA isolation and amplification from tumor sample (as determined by Argos).
2. Karnofsky performance status (KPS) score of 80-100.
3. Life expectancy of six months or greater.
4. NSCLC of any histology.
5. Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to Grade ≤ 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
6. Negative serum pregnancy test for female subjects with reproductive potential, and agreement of all male and female subjects of reproductive potential to use a reliable form of contraception during the study and for 12 weeks after the last dose of study drug.
7. Able to abstain from taking prohibited drugs, either prescription or non-prescription, during the treatment phase of the study.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
9. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Exclusion Criteria:

1. Active autoimmune disease or condition requiring chronic immunosuppressive therapy
2. Any clinically significant condition that prohibits the initiation of standard of care.
3. Malignancies within the prior three years, except for:

   * treated in situ carcinomas or non-melanoma skin cancer.
   * adequately treated early stage breast cancer.
   * superficial bladder cancer.
   * non-metastatic prostate cancer with a normal prostate-specific antigen (PSA) level.
4. History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease.
5. Clinically significant disorders or conditions including

   * cardiovascular system.
   * renal system.
   * hepatic organ system.
   * coagulation disorders.
6. Clinically significant infections, including human immunodeficiency virus (HIV), syphilis, and active hepatitis B or C.
7. Pregnant or breastfeeding.
8. Any serious medical condition or illness considered by the investigator to constitute an unwarranted high risk for investigational treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) V4.03 | 2 Years
  Safety of AGS-003-LNG for subjects who receive 1 or more doses of AGS-003-LNG in combination with standard platinum-doublet chemotherapy with or without radiation. Adverse events will be collected per CTCAE V4.03.
Immunogenicity - Generation of Cluster of Differentiation-8 (CD8)+ Cluster of Differentiation (CD28)+ memory T-cells | After 5th dose of AGS-003-LNG. Within 6 months.
  Generation of CD8+CD28+ memory T-cells against tumor associated antigens in subject receiving 5 or more doses of AGS-003-LNG.

SECONDARY OUTCOMES:
Efficacy - Overall survival | 2 Years
  While the study is not powered for efficacy Overall Survival (including median and one year survival) be analyzed as an exploratory endpoints.
Efficacy - Progression-free survival as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. | 2 Years
  While the study is not powered for efficacy, Progression Free Survival will be analyzed as an exploratory endpoint.
Efficacy - Objective response rate. The number of patients with a Complete Response or Partial Response. | 2 Years
  While the study is not powered for efficacy Objective Response Rate will be analyzed as an exploratory endpoint.
Feasibility - Number of patients with a success in the manufacture of AGS-003-LNG. | 1 Month
  AGS-003-LNG manufacturing success rate for non small cell lung cancer tumor RNA isolation from surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Luke T Nordquist, MD, Study Director — Cancer Research Network of Nebraska
Locations (1):
- Cancer Research Network of Nebraska / Oncology Associates, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No